CLINICAL TRIAL: NCT06413745
Title: A Phase II Clinical Study of SHR-A1811 in Patients With HER2-expressing/Amplified, Locally Advanced, Unresectable or Metastatic Biliary Tract Cancer (BTC) Who Have Previously Failed First or Second-line Systemic Therapy
Brief Title: Phase II Clinical Study of SHR-A1811 in Patients With HER2 Expression / Amplification of Locally Advanced Unresectable or Recurrent Metastatic Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-212
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: HER2 Expression / Amplification in Patients With Biliary Tract Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811

SUMMARY:
This study was to evaluate the efficacy and safety of SHR-A1811 in patients with locally advanced unresectable or recurrent metastatic BTC with HER2 expression / amplification who failed first-line or second-line systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old ( including both ends ), male or female ;
2. ECOG-PS score : 0 or 1;
3. Expected survival ≥ 12 weeks;
4. Subjects with locally advanced or recurrent metastatic biliary tract cancer diagnosed by histopathology or cytology are not suitable for surgical resection, transplantation or ablation;
5. Subjects who failed or intolerance after systemic chemotherapies;
6. According to the RECIST v1.1 standard, the subjects had at least one measurable lesion；
7. The main organ function is normal, in line with the program requirements ;
8. If the patient has active hepatitis B virus ( HBV ) infection : HBV-DNA must be < 500 IU / mL；
9. Consent to contraception.

Exclusion Criteria:

1. Received anti-tumor treatment such as chemotherapy, radiotherapy, immunotherapy, biotherapy or other clinical research drugs within 4 weeks before the first administration;
2. Subjects with a history or evidence of brain metastasis or meningeal metastasis ;
3. With acute or chronic uncontrolled pancreatitis or Child-Pugh liver function grade C ;
4. Severe trauma or major surgery was performed within 4 weeks before the first administration;
5. To study the severe heart disease within 6 months before the first administration ;
6. Patients with clinical symptoms and uncontrolled moderate and above pleural effusion, ascites or pericardial effusion, requiring therapeutic puncture drainage ;
7. Severe infection symptoms occurred within 2 weeks before the first administration;
8. Known hereditary or acquired bleeding and thrombotic tendency ;
9. Congenital or acquired immune defects;
10. The subjects had severe and uncontrollable concomitant diseases;
11. Cerebral infarction, pulmonary embolism or deep vein thrombosis occurred within 6 months before the first administration of the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
ORR evaluated by IRC according to RECIST v1.1 standard | About a year

SECONDARY OUTCOMES:
DoR evaluated by IRC according to RECIST v1.1 standard | About a year
DCR evaluated by IRC according to RECIST v1.1 standard | About a year
PFS evaluated by IRC according to RECIST v1.1 standard | About a year
ORR evaluated by the researchers according to the RECIST v1.1 standard | About a year
DCR evaluated by the researchers according to the RECIST v1.1 standard | About a year
DoR evaluated by the researchers according to the RECIST v1.1 standard | About a year
PFS evaluated by the researchers according to the RECIST v1.1 standard | About a year
OS | About two year
AE | About a year
SAE | About a year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided